CLINICAL TRIAL: NCT00822315
Title: Phase II Open-label Randomized Multicenter Trial to Compare the Efficacy and Safety of Two Different Doses of Raltegravir and Efavirenz, All in Combination With Tenofovir and Lamivudine, in Naive HIV-1-infected Patients Receiving Rifampin for Active Tuberculosis
Brief Title: Efficacy and Safety of 2 Raltegravir Doses in Naive HIV-1-infected Patients Receiving Rifampin for Active Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12180 REFLATE TB
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV; Tuberculosis; Pharmacokinetics; Raltegravir; France; Brazil; treatment naive
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — efavirenz; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): efavirenz
  Interventions: Drug: efavirenz
- 2 (Experimental): raltegravir 400 mg
  Interventions: Drug: raltegravir
- 3 (Experimental): raltegravir 800 mg
  Interventions: Drug: raltegravir

INTERVENTIONS:
Drug: efavirenz — tenofovir 245 mg / lamivudine 300 mg / efavirenz 600 mg
  Arms: 1
Drug: raltegravir — tenofovir 245 mg / lamivudine 300 mg / raltegravir 400 mg
  Arms: 2
Drug: raltegravir — tenofovir 245 mg / lamivudine 300 mg / raltegravir 800 mg
  Arms: 3

SUMMARY:
Raltegravir is a potent antiretroviral agent that could be used as an alternative to efavirenz in HIV-1 infected patients with tuberculosis. However due to pharmacokinetic interactions, the optimal dose of raltegravir to be used in combination with rifampin is currently unknown.

This phase II open-label randomized multicenter trial is designed to estimate the antiviral efficacy of two doses of raltegravir and one dose of efavirenz at week 24, in HIV-1 naive patients co-infected with active tuberculosis (TB) treated with rifampin.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (at least 18 years old)
* Plasma HIV RNA > 1000 copies/ml
* HIV-1-infection confirmed by ELISA and Western blot or Immunofluorescence
* ART naïve patients or
* ART for less than 3 months and more than 6 months ago ; an HIV resistance genotype at baseline showing no mutation to NNRTI and TDF or 3TC will be required
* For women of childbearing age, negative urinary test for pregnancy and to accept contraceptive methods: condom use and intra-uterine device when possible or declare no wish of pregnancy in the coming year.
* Confirmed or probable TB
* TB treatment including rifampin started since 2 to 8 weeks before randomisation
* Signed informed consent form
* For French patients, to be affiliated to the National Health Care System

Exclusion Criteria:

* HIV-2 infection (single or with HIV-1)
* Woman who is pregnant or likely to become so, is breastfeeding or refuses to use contraception
* ALT>2.5N, Hb <7g/dl, neutrophils < 750/mm3, platelet<50 000/mm3, bilirubin >5N, lipase >3N
* Creatinine clearance <60ml/min as assessed by the Cockcroft method
* Ongoing psychiatric pathology or any condition (including, but not limited to, the consumption of alcohol or drugs) which might, in the investigator's opinion, compromise the safety of treatment and/or patient compliance with the protocol
* Concomitant treatments including phenytoin or phenobarbital (compounds interacting with UGT1A1)
* Prior TB with a Mycobacterium tuberculosis strain resistant to rifampin
* TB treatment started for more than 8 weeks before randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Virologic success, using Time to Loss of Virologic Response (TLOVR) algorithm: -Plasma HIV RNA below 50 copies/ml at week 20, confirmed at week 24 -Absence of permanent treatment discontinuation -Absence of death -Still follow-up at week 24 | 24 weeks

SECONDARY OUTCOMES:
Proportion of patients with virologic response with the following definitions: - Plasma HIV RNA <50 copies/ml at week 24 - Rate of strategy discontinuation and treatment changes - Proportion of death - Proportion of patients loss to follow-up | 24 weeks
Proportion of patients with virologic response with the following definitions: o Plasma HIV RNA <50 copies/ml o Plasma HIV RNA <400 copies/ml | 24 and 48 weeks
Evolution in HIV RNA and HIV DNA (total and 2 LTR circular) from baseline to week 48 | 48 weeks
Rate of viral resistance mutations in the plasma at the time of virologic failure and in comparison with HIV-RNA mutations at W0 | At the time of virologic failure
Evolution of CD4 cell counts from baseline to week 48 | 48 weeks
Frequency, type and time to a new AIDS-defining event or death | Through out the trial
Frequency, type, time to grade 3 or 4 adverse event | Through out the trial
Rate of success of TB treatment | 48 weeks
Anti-TB resistance rate | 48 weeks
Evolution of raltegravir and efavirenz trough concentration | Through out the trial

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Grinsztejn, MD, Study Chair — Fiocruz, Rio de Janiero, Brazil; Jean-Michel Molina, MD, Study Chair — Hôpital Saint-Louis, Paris, France
Locations (9):
- Brazil (6):
  - Hospital Genral de Nova Iguaçu, Nova Iguaçu
  - Hospital Nossa Senhora da Coceiçao, Porto Alegre
  - Hospital Sanatorio Pertenon, Porto Alegre
  - Ipec/Fiocruz, Rio de Janeiro
  - Hospitral Universitario Pr Edgar Santos, Salvador
  - STD/AIDS department, São Paulo
- France (3):
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Louis, Paris
  - CHI Villeneuve Saint Georges, Villeneuve-Saint-Georges

REFERENCES:
- [Derived] Grinsztejn B, De Castro N, Arnold V, Veloso VG, Morgado M, Pilotto JH, Brites C, Madruga JV, Barcellos NT, Santos BR, Vorsatz C, Fagard C, Santini-Oliveira M, Patey O, Delaugerre C, Chene G, Molina JM; ANRS 12 180 Reflate TB study group. Raltegravir for the treatment of patients co-infected with HIV and tuberculosis (ANRS 12 180 Reflate TB): a multicentre, phase 2, non-comparative, open-label, randomised trial. Lancet Infect Dis. 2014 Jun;14(6):459-67. doi: 10.1016/S1473-3099(14)70711-X. Epub 2014 Apr 9. PMID 24726095